CLINICAL TRIAL: NCT04899154
Title: MEDIBIOTE 3: Analysis of Intestinal Microbiota as a Predictor of Response to Treatment of Spondyloarthritis With Biotherapy
Brief Title: Analysis of Intestinal Microbiota as a Predictor of Response to Treatment of Spondyloarthritis With Biotherapy
Acronym: MEDIBIOTE 3
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hôpital Européen Marseille (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2018-A03050-55
Record Dates: First submitted 2021-05-19; First posted 2021-05-24 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Spondyloarthritis
MeSH Terms: conditions — Spondylarthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients with spondyloarthritis (Spa) (Experimental)
  Interventions: Other: stool sampling
- Healthy subjects (Experimental)
  Interventions: Other: stool sampling

INTERVENTIONS:
Other: stool sampling — Participants will provide two stool samples: one collected the day of inclusion and a second, four months later after anti-TNF α or anti- IL-17 (interleukin-17) treatment initiation.
  Arms: Patients with spondyloarthritis (Spa)
Other: stool sampling — Participants will provide one stool sample at inclusion
  Arms: Healthy subjects

SUMMARY:
Spondyloarthritis (SpA) is a group of inflammatory rheumatic disorders that mainly manifested by inflammatory pain of the spine, pelvis and sometimes limbs. Classically, SpA has been classified into several subtypes, such as ankylosing spondylitis (AS), psoriatic arthritis (PsA), inflammatory bowel disease (IBD)-associated.

Several studies have shown specific changes in the gut microbiota during SpA. A recent, uncontrolled study suggested that the therapeutic response to anti-TNFα (Tumor Necrosis Factor) therapy could be predicted by analysis of the gut microbiota.

The purpose of the study MEDIBIOTE 3 is to confirm that in SpA, the composition of the intestinal microbiota at the initiation of treatment is predictive of the response to treatment with biotherapy (anti-TNFα / anti-IL17).

ELIGIBILITY:
Inclusion Criteria:

For patient with spondyloarthritis:

* Diagnosed for spondyloarthritis or pure axial or axial type psoriatic rheumatism according to Assessment of Spondyloarthritis International Society (ASAS) criteria.
* Requiring treatment with anti-TNFα or anti- IL-17 according to the treatment recommendations of the French Society of Rheumatology (SFR)
* patient not previously treated with biotherapy
* Aged ≥ 18 years
* Having given free and informed written consent
* Being affiliated to the center national security system social

For control Subject:

* Healthy volunteers without diagnosis of spondyloarthritis or any other chronic disease.
* Aged ≥ 18 years
* Having given free and informed written consent
* Being affiliated with or benefiting from a social security scheme.

Exclusion Criteria:

* Persons treated with antibiotics, probiotics, prebiotics or any other treatment that may disrupt the gut microbiota within one month before stool sampling.
* Association with another chronic pathology

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2019-07-16 (Actual); Primary Completion 2026-05-15 (Estimated); Study Completion 2026-05-15 (Estimated)

PRIMARY OUTCOMES:
Variability in the qualitative and quantitative composition of intestinal microbiota in patients responding to biotherapy compared to the group of non-responding patients | 18 Months

SECONDARY OUTCOMES:
Differences on intestinal microbiota composition (qualitative and quantitative) of patients with Spa versus healthy controls. | 18 Months

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Européen Marseille, Marseille, France

IPD SHARING:
Plan to Share IPD: No